CLINICAL TRIAL: NCT01104987
Title: Treatment With Alendronate in Patients With Ankylosing Spondylitis (AS), an Open Label Prospective Trial
Brief Title: Treatment With Alendronate in Patients With Ankylosing Spondylitis (AS)
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 20090618
Record Dates: First submitted 2010-04-13; First posted 2010-04-16 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Ankylosing Spondylitis; Osteoporosis
Keywords: Ankylosing spondylitis; spondarthritis; Osteoporosis; Bone mineral density; Dual energy x-ray absorptiometry; Quantitative computed tomography
MeSH Terms: conditions — Spondylitis, Ankylosing; Osteoporosis; Spondylarthritis | interventions — Alendronate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- alendronate: A cross sectional study assessing the prevalence of osteoporosis and vertebral fractures in AS has been conducted during the spring in 2009. Patients with osteoporosis that fulfilled the inclusion criteria and did not have any exclusion criteria for the present trial were asked to join this study.
  Interventions: Drug: alendronate

INTERVENTIONS:
Drug: alendronate — One tablet of alendronate à 70 mg once a week during two years.

SUMMARY:
This prospective study will assess the effects of treatment with alendronate in osteoporotic patients with ankylosing spondylitis.

Primary objectives:

* To investigate if alendronate effect bone mineral density (BMD) assessed by dual energy x-ray absorptiometry (DXA) in lumbar spine, hip and distal forearm and assessed by quantitative computed tomography (QCT) in lumbar spine and by Xtreme CT in radius and tibia.

Secondary objectives:

* To investigate if alendronate effects markers of bone remodeling
* To investigate if alendronate influences disease activity (BASDAI), spinal function (BASFI), spinal movement (BASMI) and health related quality of life (SF-36).

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a common inflammatory rheumatic disease with a prevalence of 0.5-1.0%. Men are more commonly affected by the disease as compared to women, ratio 2.6-4:1. Pain in the back is a frequent symptom of debut. This pain is often associated with sacroilitis. In later stages also the lumbar, thoracic and cervical spine are hit by the disease. Peripheral joints, eyes, heart, lungs and urinary tract may also be influenced.

The risk of osteoporosis is increased in AS. However, this field has not yet been significantly studied probably due to several reasons such as the predominance of men with the disease and men are more seldom investigated for osteoporosis compared to women. When AS progresses syndesmophytes of the spine are developed which makes it difficult to assess bone mineral density (BMD) correctly with the conventional method, dual energy x-ray absorptiometry (DXA). Fractures in the spine are easy to foreseen since the pain of the patient might be misjudged to be related to increased disease activity. Fractures are also overlooked in radiographs in AS. AS is associated with both increased bone formation and increased bone resorption. The bone remodeling process in the spine renders the spine less flexible and stiffer and as a consequence also a quite small trauma may result in a fracture. These fractures are often instable risking injuring the spinal cord and nerves.

Treatment with bisphosphonates in AS have indicated an anti-inflammatory effect. The effects of treatment with bisphosphonate on BMD assessed by DXA, QCT and Xtreme CT in AS has not yet been fully investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill diagnostic criteria of ankylosing spondylitis, 1984 New York
2. Patients should previously have been included in the observational trial, "Clinical study of osteoporosis in ankylosing spondylitis".
3. Patients should not have changed treatment with any biologics the past 4 months.
4. Patients on glucocorticosteroids should not have changed the dose the last 4 months.
5. BMD with a T-score ≤ -2,5 SD assessed by DXA in lumbar spine and/or hip (total hip and/or neck).
6. BMD with a T-score ≤ -2,0 SD assessed by DXA in lumbar spine and/or hip (total hip and/or neck) and presence of any vertebral fracture, hip fracture or peripheral fragility fracture.
7. BMD with a T-score ≤ - 1,0 SD assessed by DXA in lumbar spine and/or hip (total hip and/or neck) in patients on oral glucocorticosteroids

Exclusion criteria:

1. Ongoing treatment with any bisphosphonate.
2. Ongoing treatment with any sex-hormone.
3. Renal insufficiency, creatinine clearance < 35 ml/min
4. Difficulties in swallowing and/or acute illness in the upper gastro-intestinal canal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AS and osteoporosis.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 2 years
  The effect on bone mineral density (BMD) assessed by dual energy x-ray absorptiometry (DXA) in lumbar spine, hip and distal forearm and assessed by quantitative computed tomography (QCT) in lumbar spine and by Xtreme CT in radius and tibia by treatment with alendronate.

SECONDARY OUTCOMES:
Markers of bone remodeling | 2 years
  To investigate the effects on serum markers of bone remodeling by treatment with alendronate.
Disease activity | 2 years
  To investigate if alendronate influences disease activity measured by the validated instrument BASDAI.
Spinal function | 2 years
  To investigate if alendronate influences spinal function measured by the validated instrument BASFI.
Spinal movement | 2 years
  To investigate if alendronate influences spinal movement measured by the validated instrument BASMI.
Health related quality of life | 2 years
  To investigate if alendronate influences health related quality of life measured by the validated instrument SF-36.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Forsblad d'Elia, MD, PhD, Principal Investigator — Sahlgrenska Academy at University of Gothenburg, Department of Rheumatology and Inflammation Research
Locations (1):
- Department of Rheumatology, Sahlgrenska University Hospital, Gothenburg, Sweden